CLINICAL TRIAL: NCT01211587
Title: A Double-blind, Randomized, Placebo-controlled, Parallel-group Phase II Study to Explore the Potential Beneficial Effects of Safinamide on Cognition in Non-demented Patients With Idiopathic Parkinson's Disease (PD) and Cognitive Impairment
Brief Title: A Trial to Explore the Potential Benefit of Safinamide on Cognitive Impairment Associated With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMR701165-024
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2012-06

CONDITIONS: Parkinson's Disease With Cognitive Impairments
Keywords: Parkinson's Disease; Cognition; Safinamide; Phase 2; Non-demented patients; Levodopa; Dopamine agonist
MeSH Terms: conditions — Parkinson Disease | interventions — safinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 100mg safinamide (Experimental): Two 50mg tablets of safinamide once per day for 12 weeks (weeks 1-12) Open Label part: Two 50mg tablets of safinamide once per day for 12 weeks (week 13-24)
  Interventions: Drug: safinamide
- Placebo (Placebo Comparator): Two 50mg tablets of placebo once per day for 12 weeks (weeks 1-12) Open Label part: Two 50mg tablets of safinamide once per day for 12 weeks (week 13-24)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: safinamide — Safinamide will be provided in tablets equivalent to 50 mg in blisters. After randomization, patients receiving safinamide will take two 50 mg tablets once per day for 12 weeks (weeks 1-12). During the open label phase, patients will receive 100mg of safinamide once per day (two 50 mg tablets) for 12 weeks (weeks 13-24).
  Arms: 100mg safinamide
Drug: placebo — Identical placebo tablets will be provided in blisters. After randomization, patients receiving placebo will take two tablets once per day for 12 weeks (weeks 1-12). During the open label phase, patients will receive 100mg of safinamide once per day (two 50 mg tablets) for 12 weeks (weeks 13-24).
  Arms: Placebo

SUMMARY:
The purpose of this research trial is to determine if safinamide (experimental drug) can improve cognition in cognitively impaired but non-demented Parkinson's disease patients. The word "experimental" means the trial drug is not approved by Health Authorities (government authorities) and is still being tested for safety and effectiveness.

Approximately one hundred (100) patients will participate in this research trial. The research trial will be conducted in approximately thirty (30) medical centers in the following countries: Argentina, Canada, Italy, Peru, South Africa, Spain and USA. The research trial will last until June 2012.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients (aged 45 to 80 years inclusive)
* Diagnosis of idiopathic Parkinson's Disease (PD) according to the UK PDS Brain Bank Criteria and a Hoehn and Yahr Stage of I to III (mild to moderate motor severity) at Screening. The diagnosis will be based on medical history and neurological examination
* Subjects and informants must report cognitive impairment in at least one cognitive domain on the PD Cognitive Questionnaire (PD-CQ).
* Cognitive impairment confirmed by a total score equal to- or below 26 on the Montreal Cognitive Assessment (MoCA)
* Be able to speak, read, and write in the language in which the tests are written and must be able to perform all the assessments in this language
* Receiving treatment with dopaminergic therapy (dopamine agonist and/or levodopa at a stable dose for at least four weeks prior to Screening and for the duration of the study)
* Understand and sign the appropriate approved Informed Consent Form(s), one for the study (mandatory) and one for the pharmacogenetic evaluation (optional)

Exclusion Criteria:

* Any indication of forms of Parkinsonism other than idiopathic PD
* Diagnosis of PD Dementia (probable, possible) according to the Clinical Diagnostic Criteria for Dementia Associated with PD
* Diagnosis of Dementia with Lewy Bodies according to the McKeith criteria.
* Subjects with any clinically significant DSM-IV-TR Axis I Disorders including major depression and severe anxiety; current diagnosis of substance abuse or history of alcohol or drug abuse for 3 months prior to Visit 1 (Screening)
* Mental/physical/social condition which could preclude performing efficacy or safety assessments
* Severe white matter disease, multiple lacunar infarcts, or signs of significant vascular changes on Magnetic Resonance Imaging (MRI)
* Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer(ed) from such
* Current history of severe dizziness or fainting on standing, due to postural hypotension
* Second- or third-degree atrioventricular block or sick sinus syndrome, uncontrolled atrial fibrillation, severe or unstable angina, congestive heart failure, myocardial infarction in the three months prior to Visit 1 (Screening), or significant electrocardiogram (ECG) abnormality, including heart-rate corrected interval QT (QTC) > 450 milliseconds (males) or > 470 milliseconds (females), with QTC based on the Bazett's correction method
* Known diagnosis of human immunodeficiency virus (HIV) infection, positive results on tests for hepatitis B or C antibodies, or on tests for hepatitis B surface antigen (unless vaccinated)
* Neoplastic disease, either currently active or in remission for less than 1 year
* Clinically significant or unstable gastrointestinal, renal, hepatic, endocrine, pulmonary, or cardiovascular disease, including not well controlled hypertension, asthma, chronic obstructive pulmonary disease, and Type 1 diabetes that would, in the opinion of the Investigator, preclude participation to the study
* Any clinically relevant abnormality, either on medical history, physical and neurological examination, ECG, or by diagnostic laboratory tests that, in the opinion of the Investigator, could hinder participation to the study
* Currently experiencing end-of-dose wearing-off or on-off phenomena, disabling peak dose- or biphasic dyskinesia, or unpredictable or widely swinging fluctuations
* Any medical conditions and/or taking concomitant medications that could put them at risk, interfere with study evaluations, or prevent meeting the requirements of the study
* Currently participating to another clinical trial or who participated in a previous clinical trial within 30 days prior to Visit 1 (Screening) or who received any investigational product within 30 days or five half-lives, whichever was longer, prior to Visit 1 (Screening)
* Previously treated with safinamide
* Clinically significant hypertension or contraindications or hypersensitivity to monoamine oxidase-Type B (MAO-B) inhibitors
* Anticholinergic medication and/or amantadine within 4 weeks prior to the Screening visit
* Opioids (e.g., tramadol and meperidine derivatives) or MAO inhibitors (e.g., selegiline) within 8 weeks prior to Visit 1 (Screening) Dextromethorphan will be allowed to treat cough. One tricyclic- or tetracyclic antidepressant or trazodone will be permitted if taken at bedtime at a low dose as a sleeping aid
* Acetylcholinesterase inhibitors or memantine within 4 weeks before start of the study treatment or requiring these medications during the treatment period
* Depot neuroleptic during the study or within 1 injection cycle or oral neuroleptics (stable dose of quetiapine less than 100 mg/day for 8 weeks prior to Visit 1 will be allowed) within 4 weeks prior to Visit 1 (Screening)
* Drug that has hepatotoxic potential (e.g., tamoxifen) within 4 weeks prior to Visit 1 (Screening), or radiation therapy, or a drug with cytotoxic potential (e.g., chemotherapy) within 1 year prior to the Screening visit.
* Subjects who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study
* Women who are pregnant, lactating, or who are attempting to conceive
* Women of childbearing potential not willing to use an adequate contraceptive method (unless surgically sterilized) for 4 weeks prior to, during, and 4 weeks after the last dose of trial medication
* Clinically significant ophthalmologic abnormality such as patients with albinism, family history of hereditary retinal disease, progressive and/or severe diminution of corrected visual acuity, retinitis pigmentosa, any active retinopathy or ocular inflammation (uveitis), or progressive, severe diabetic retinopathy
* Known hypersensitivity to the trial treatment(s), including placebo or other comparator drug(s)
* Legal incapacity or limited legal capacity

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Parkinson's Disease Cognitive Rating Scale (PD-CRS) | 12 weeks
  Total score reduction in the PD-CRS at 12 weeks compared to the Baseline. The PD-CRS detects early cognitive impairment in Parkinson's disease. It is composed of 2 scales, the subcortical scale (items 1, 3, 4, 5, 7, 8, 9) and the cortical scale (items 2, 6). The total score of the subcortical scale is from 0 to 114. The total score of the cortical scale is from 0 to 20. The PD-CRS Total score represents the sum of scores on the cortical and subcortical scales. It ranges from 0 to 134. The more points, the less the impairment.

SECONDARY OUTCOMES:
PD-CRS subscale scores | 6 weeks
  The PD-CRS detects early cognitive impairment in Parkinson's disease. It is composed of 2 scales, the subcortical scale (items 1, 3, 4, 5, 7, 8, 9) and the cortical scale (items 2, 6). The total score of the subcortical scale is from 0 to 114. The total score of the cortical scale is from 0 to 20. The PD-CRS Total score represents the sum of scores on the cortical and subcortical scales. It ranges from 0 to 134. The more points, the less the impairment.
PD-CRS subscale scores | 24 weeks
  The PD-CRS detects early cognitive impairment in Parkinson's disease. It is composed of 2 scales, the subcortical scale (items 1, 3, 4, 5, 7, 8, 9) and the cortical scale (items 2, 6). The total score of the subcortical scale is from 0 to 114. The total score of the cortical scale is from 0 to 20. The PD-CRS Total score represents the sum of scores on the cortical and subcortical scales. It ranges from 0 to 134. The more points, the less the impairment.
PD-CRS total score | 24 weeks
  The PD-CRS detects early cognitive impairment in Parkinson's disease. It is composed of 2 scales, the subcortical scale (items 1, 3, 4, 5, 7, 8, 9) and the cortical scale (items 2, 6). The total score of the subcortical scale is from 0 to 114. The total score of the cortical scale is from 0 to 20. The PD-CRS Total score represents the sum of scores on the cortical and subcortical scales. It ranges from 0 to 134. The more points, the less the impairment.
Dementia Rating Scale - 2 (DRS-2) total score | 12 weeks
  DRS-2 will provide a general measure of cognitive ability in PD subjects. It has thus been chosen as a tool to compare cognitive performance in PD across different trials. Administered at Baseline, Week 12 and Week 24. The DRS-2 consists of 36 tasks divided into 5 subscales (Attention, Initiation/Perseveration, Construction, Conceptualization, and Memory). The maximum score on each subscale is as follows: Attention = 37; Initiation/Perseveration = 37; Construction = 6; Conceptualization = 39, Memory = 25. The DRS-2 total score = 144 (the more points, the less the impairment).
DRS-2 total score | 24 weeks
  DRS-2 will provide a general measure of cognitive ability in PD subjects. It has thus been chosen as a tool to compare cognitive performance in PD across different trials. Administered at Baseline, Week 12 and Week 24. The DRS-2 consists of 36 tasks divided into 5 subscales (Attention, Initiation/Perseveration, Construction, Conceptualization, and Memory). The maximum score on each subscale is as follows: Attention = 37; Initiation/Perseveration = 37; Construction = 6; Conceptualization = 39, Memory = 25. The DRS-2 total score = 144 (the more points, the less the impairment).
DRS-2 subscale scores | 12 weeks
  DRS-2 will provide a general measure of cognitive ability in PD subjects. It has thus been chosen as a tool to compare cognitive performance in PD across different trials. Administered at Baseline, Week 12 and Week 24. The DRS-2 consists of 36 tasks divided into 5 subscales (Attention, Initiation/Perseveration, Construction, Conceptualization, and Memory). The maximum score on each subscale is as follows: Attention = 37; Initiation/Perseveration = 37; Construction = 6; Conceptualization = 39, Memory = 25. The DRS-2 total score = 144 (the more points, the less the impairment).
DRS-2 subscale scores | 24 weeks
  DRS-2 will provide a general measure of cognitive ability in PD subjects. It has thus been chosen as a tool to compare cognitive performance in PD across different trials. Administered at Baseline, Week 12 and Week 24. The DRS-2 consists of 36 tasks divided into 5 subscales (Attention, Initiation/Perseveration, Construction, Conceptualization, and Memory). The maximum score on each subscale is as follows: Attention = 37; Initiation/Perseveration = 37; Construction = 6; Conceptualization = 39, Memory = 25. The DRS-2 total score = 144 (the more points, the less the impairment).
Clinical Global Impression (CGI) Change in Cognitive Dysfunction (CGI-C Cognition) | 6 weeks
  CGI is a clinician-rated instrument assessing the severity (CGI-S) and the improvement/change (CGI-C) of PD over time scale. The original scale has been adapted to assess the severity of cognitive dysfunctions and the change/improvement in cognitive dysfunctions over time. Rating will be based on a Likert-type scale (0 = Not assessed, 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse). The maximum score on the scale is 7. The CGI-C Cognition will be administered at 6 weeks, 12 weeks, and 24 weeks.
CGI-C Cognition | 24 weeks
  CGI is a clinician-rated instrument assessing the severity and the improvement/change of PD over time scale. The original scale has been adapted to assess the severity of cognitive dysfunctions and the change/improvement in cognitive dysfunctions over time. Rating will be based on a Likert-type scale (0 = Not assessed, 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse). The maximum score on the scale is 7. The CGI-C Cognition will be administered at 6 weeks, 12 weeks, and 24 weeks.
CGI-Severity in Cognitive Dysfunction (CGI-S Cognition) | 6 weeks
  CGI is a clinician-rated instrument assessing the severity and the improvement/change of PD over time scale. The original scale has been adapted to assess the severity of cognitive dysfunctions and the change/improvement in cognitive dysfunctions over time. Rating will be based on a Likert-type scale (0 = Not assessed, 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse). The maximum score on the scale is 7. The CGI-S Cognition will be administered at Baseline, 6 weeks, 12 weeks, and 24 weeks.
CGI-S Cognition | 24 weeks
  CGI is a clinician-rated instrument assessing the severity and the improvement/change of PD over time scale. The original scale has been adapted to assess the severity of cognitive dysfunctions and the change/improvement in cognitive dysfunctions over time. Rating will be based on a Likert-type scale (0 = Not assessed, 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse). The maximum score on the scale is 7. The CGI-S Cognition will be administered at Baseline, 6 weeks, 12 weeks, and 24 weeks.
Patient's Clinical Global Impression of Change in Cognitive (PCGI-C Cognition) | 6 weeks
  CGI is a clinician-rated instrument assessing the severity and the improvement/change of PD over time scale. Subjects will be asked to rate their own change in cognition using the CGI-C. This rating will be the PCGI-C Cognition. Rating will be based on a Likert-type scale (0 = Not assessed, 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse). The maximum score on the scales is 7. The Patient's Change in Cognitive Dysfunction (PCGI-C) will be administered at 6 weeks, 12 weeks, and 24 weeks.
PCGI-C Cognition | 24 weeks
  CGI is a clinician-rated instrument assessing the severity and the improvement/change of PD over time scale. Subjects will be asked to rate their own change in cognition using the CGI-C. This rating will be the PCGI-C Cognition. Rating will be based on a Likert-type scale (0 = Not assessed, 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse). The maximum score on the scales is 7. The Patient's Change in Cognitive Dysfunction (PCGI-C) will be administered at 6 weeks, 12 weeks, and 24 weeks.
Grid-Hamilton Depression Rating Scale (Grid-HAMD) | 6 weeks
  Grid-HAMD uses a grid-like structure to separates the frequency from the intensity of a symptom. The 17 items of the scale are rated on a 5-point (0-4) or 3-point (0-2) scale. Items using the 5-point scale are rated as 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), or 4 (very severe). Items using the 3-point scale are rated as 0 (absent), 1 (probable), or 2 (definite). The higher the score, the greater the depression. The scale will be administered at Baseline, 6 weeks, 12 weeks, and 24 weeks.
Grid-HAMD | 24 weeks
  Grid-HAMD uses a grid-like structure to separates the frequency from the intensity of a symptom. The 17 items of the scale are rated on a 5-point (0-4) or 3-point (0-2) scale. Items using the 5-point scale are rated as 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), or 4 (very severe). Items using the 3-point scale are rated as 0 (absent), 1 (probable), or 2 (definite). The higher the score, the greater the depression. The scale will be administered at Baseline, 6 weeks, 12 weeks, and 24 weeks.
Parkinson's Disease Sleep Scale (PDSS) | 6 weeks
  PDSS addresses commonly reported symptoms associated with sleep disturbance: Overall quality of night's sleep (item 1); Sleep onset and maintenance insomnia (items 2&3); Nocturnal restlessness (items 4&5); Nocturnal psychosis (items 6&7); Nocturia (items 8&9); Nocturnal motor symptoms (items 10-13); Sleep refreshment (item 14); Daytime dozing (item 15). Scores for each item range from 0 (symptom severe & always experienced) to 10 (symptom-free). The maximum cumulative score is 150 (subject is free of all symptoms). The PDSS will be administered at Baseline, 6 weeks, 12 weeks, and 24 weeks.
PDSS | 24 weeks
  PDSS addresses commonly reported symptoms associated with sleep disturbance: Overall quality of night's sleep (item 1); Sleep onset and maintenance insomnia (items 2&3); Nocturnal restlessness (items 4&5); Nocturnal psychosis (items 6&7); Nocturia (items 8&9); Nocturnal motor symptoms (items 10-13); Sleep refreshment (item 14); Daytime dozing (item 15). Scores for each item range from 0 (symptom severe & always experienced) to 10 (symptom-free). The maximum cumulative score is 150 (subject is free of all symptoms). The PDSS will be administered at Baseline, 6 weeks, 12 weeks, and 24 weeks.
Apathy Scale (AS) | 6 weeks
  AS is a tool to measure severity of apathy in PD subjects. It consists of 14 questions that are to be answered on a four-point Likert scale. The maximum score is 42 with a low and high apathy cut-off score of 14. The AS will be administered at Baseline, 6 weeks, 12 weeks, and 24 weeks.
AS | 24 weeks
  AS is a tool to measure severity of apathy in PD subjects. It consists of 14 questions that are to be answered on a four-point Likert scale. The maximum score is 42 with a low and high apathy cut-off score of 14. The AS will be administered at Baseline, 6 weeks, 12 weeks, and 24 weeks.
CGI-C Cognition | 12 weeks
  CGI is a clinician-rated instrument assessing the severity (CGI-S) and the improvement/change (CGI-C) of PD over time scale. The original scale has been adapted to assess the severity of cognitive dysfunctions and the change/improvement in cognitive dysfunctions over time. Rating will be based on a Likert-type scale (0 = Not assessed, 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse). The maximum score on the scale is 7. The CGI-C Cognition will be administered at 6 weeks, 12 weeks, and 24 weeks.
CGI-S Cognition | 12 weeks
  CGI is a clinician-rated instrument assessing the severity and the improvement/change of PD over time scale. The original scale has been adapted to assess the severity of cognitive dysfunctions and the change/improvement in cognitive dysfunctions over time. Rating will be based on a Likert-type scale (0 = Not assessed, 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse). The maximum score on the scale is 7. The CGI-S Cognition will be administered at Baseline, 6 weeks, 12 weeks, and 24 weeks.
PCGI-C Cognition | 12 weeks
  CGI is a clinician-rated instrument assessing the severity and the improvement/change of PD over time scale. Subjects will be asked to rate their own change in cognition using the CGI-C. This rating will be the PCGI-C Cognition. Rating will be based on a Likert-type scale (0 = Not assessed, 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse). The maximum score on the scales is 7. The Patient's Change in Cognitive Dysfunction (PCGI-C) will be administered at 6 weeks, 12 weeks, and 24 weeks.
Grid-HAMD | 12 weeks
  Grid-HAMD uses a grid-like structure to separates the frequency from the intensity of a symptom. The 17 items of the scale are rated on a 5-point (0-4) or 3-point (0-2) scale. Items using the 5-point scale are rated as 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), or 4 (very severe). Items using the 3-point scale are rated as 0 (absent), 1 (probable), or 2 (definite). The higher the score, the greater the depression. The scale will be administered at Baseline, 6 weeks, 12 weeks, and 24 weeks.
PDSS | 12 weeks
  PDSS addresses commonly reported symptoms associated with sleep disturbance: Overall quality of night's sleep (item 1); Sleep onset and maintenance insomnia (items 2&3); Nocturnal restlessness (items 4&5); Nocturnal psychosis (items 6&7); Nocturia (items 8&9); Nocturnal motor symptoms (items 10-13); Sleep refreshment (item 14); Daytime dozing (item 15). Scores for each item range from 0 (symptom severe & always experienced) to 10 (symptom-free). The maximum cumulative score is 150 (subject is free of all symptoms). The PDSS will be administered at Baseline, 6 weeks, 12 weeks, and 24 weeks.
AS | 12 weeks
  AS is a tool to measure severity of apathy in PD subjects. It consists of 14 questions that are to be answered on a four-point Likert scale. The maximum score is 42 with a low and high apathy cut-off score of 14. The AS will be administered at Baseline, 6 weeks, 12 weeks, and 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Willmer, MD, FRCPC, Study Director — Merck Serono S.A., Geneva
Locations (15):
- United States (9):
  - The Parkinson's Institute, Sunnyvale, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - US Medical Information Located in, Rockland, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - Baylor College of Medicine Parkinson's Disease Center and Movement Disorders Clinic, Houston, Texas
- Spain (6):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital De La Santa Creui Sant Pau, Barcelona
  - Hospital General de Catalunya, Barcelona
  - USP Institut Universitari Dexeus, Barcelona
  - Hosptial General Univ Gregorio Maranon, Madrid
  - Hospital Mutual de Terrassa, Terrassa - Barcelona